CLINICAL TRIAL: NCT04440722
Title: Prospective Observational Study and Biobank in All Persons Referred to Center of Gender Identity Odense University Hospital (CKIO)/Body Identity Clinic
Brief Title: Prospective Observational Study and Biobank CKIO
Status: Suspended | Type: Observational
Why Stopped: replaced by other study
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, Consultat, Dr Med, professor, Odense University Hospital
Other Study IDs: BICTX02
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Transgender

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine, hair
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Transgender individuals: All transgender individuals referred to center of gender identity Odense

SUMMARY:
Prospective observational study and biobank in all persons referred to CKIO

* Patient involvement and quality of life
* Population characteristics regarding hormone levels, safety parameters and clinical outcome before and after gender affirming hormone treatment.

DETAILED DESCRIPTION:
This is a prospective observational cohort study including all patients referred to the Center of Gender Identity Odense. The purpose is to follow patients yearly to observe patient reported outcomes and control the quality and effects of the clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* All Individuals with gender dysforia who are referred to Center of Gender Identity Odense
* Age 18+

Exclusion Criteria:

°There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred til CKIO
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2040-08-01 (Estimated); Study Completion 2040-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcomes (PRO) | Every 52 weeks
  Questionnaires
Hormone levels | Every 52 weeks
  Blood samples
Safety parameters | Every 52 weeks
  Blood samples

SECONDARY OUTCOMES:
Blood pressure | Every 52 weeks
  Blood pressure measured in a sitting position
Body mass index | Every 52 weeks
  Body mass index calculated from height an weight
Body weight | Every 52 weeks
  Body weight measured on a scale in kilogram
Hair cortisol | Every 52 weeks
  Hair samples 3 mm thick from the back of the head
Cortisol metabolism | Every 52 weeks
  24 hour urine samples
Spirometry | Every 52 weeks
  Forced vital capacity is measured by a spirometer

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided